CLINICAL TRIAL: NCT02802787
Title: Implementation and Evaluation of an Activity Based Program to Improve Quality of Life Outcomes in Women Diagnosed With Cancer
Brief Title: Implementation and Evaluation of an Activity Program to Improve Quality of Life Outcomes in Women Diagnosed With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: University of the Sciences in Philadelphia (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 776234-4
Record Dates: First submitted 2016-06-02; First posted 2016-06-16 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Cancer
Keywords: Quality of life; Occupation; Pain; Fatigue
MeSH Terms: conditions — Neoplasms; Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Camp Discovery (Experimental): One week activity based camp
  Interventions: Other: Camp Discovery

INTERVENTIONS:
Other: Camp Discovery — Activities will include physical, social, emotional, sensory and spiritual activities.

SUMMARY:
Implementation and Evaluation of an Activity Based Program to Improve Quality of Life, Pain and Fatigue Outcomes in Women Diagnosed With Cancer. Demonstrate improved life satisfaction, decreased pain and decreased fatigue (with evidenced gathered at three consecutive periods Quality of Life, Pain and Fatigue surveys).

DETAILED DESCRIPTION:
This research study will focus on developing and implementing two one-week activity camps in the summer of 2016 for women diagnosed with cancer. One camp will be held in West Philadelphia and another in Camden, New Jersey, both of which have been identified as underserved areas for health access. The focus of this programming is to allow women to engage in activities they may not be engaged in since the diagnosis of cancer and to provide them with opportunities to socially interact and communicate with individuals who may have encountered the same difficulties as them. Quality of life, pain and fatigue information will be collected before, during and after implementation of the activity program. The main objective is to demonstrate improved life satisfaction, decreased pain and decreased fatigue (with evidenced gathered at three consecutive periods and geographical locations through Quality of Life, Pain and Fatigue surveys). The intended sample size is 57 women.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with cancer
* Age of 21 of older
* Clearance from their MD to participate in the activity program

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure Scores at Day1, Day 5 and Week 6 | Day 1, Day 5 and week 6
  Individualized, client-centered measure designed for use by occupational therapists to detect change in a client's self-perception of occupational performance and satisfaction over time

SECONDARY OUTCOMES:
Change in Brief Pain Inventory | Day 1, Day 5, and week 6
  Pain assessment that measures level of pain will be reported for Day 1, Day 5, and Week 6
Change in Brief Fatigue Inventory | Day 1, Day 5, and week 6
  Fatigue assessment that measures level of Fatigue will be reported for Day 1, Day 5, and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle J Mendonca, PhD, Principal Investigator — Temple University
Locations (1):
- Community in Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No